CLINICAL TRIAL: NCT04047797
Title: A Phase 2 Study of Ixazomib and Rituximab in Bruton Tyrosine Kinase Inhibitor Resistant Mantle Cell Lymphoma
Brief Title: Ixazomib and Rituximab in Treating Patients With Relapsed or Refractory Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively Complete 75%<Participants
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1090; NCI-2019-04857 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-1090 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ixazomib; MLN2238; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ixazomib, rituximab) (Experimental): Patients receive ixazomib by mouth on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV over 4-8 hours on days 1, 8, 15, and 22 of cycle 1. Beginning in cycle 3, patients receive rituximab Intravenous over 4-8 hours on day 1. Treatment repeats every 28 days up to cycle 12 in the absence of disease progression or unacceptable toxicity. Patients benefiting from treatment may continue to receive ixazomib indefinitely in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib; Drug: Ixazomib Citrate; Biological: Rituximab

INTERVENTIONS:
Drug: Ixazomib — Given by mouth
  Other Names: MLN-2238; MLN2238
Drug: Ixazomib Citrate — Given by mouth
  Other Names: MLN-9708; MLN9708; Ninlaro
Biological: Rituximab — Given Intravenous
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima

SUMMARY:
This phase II trial studies how well ixazomib and rituximab work in treating patients with mantle cell lymphoma that has come back (relapsed) or does not respond (refractory) to BTK inhibitor treatment. Ixazomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with rituximab may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving ixazomib and rituximab may work better in treating patients with mantle cell lymphoma compared to rituximab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the complete remission rate of Bruton's tyrosine kinase (BTK) inhibitor refractory mantle cell lymphoma (MCL) patients with ixazomib citrate (ixazomib) and rituximab at 16 weeks of therapy.

SECONDARY OBJECTIVES:

I. To evaluate overall response rate (ORR) assessed by Lugano criteria. II. To evaluate progression free survival (PFS) and overall survival (OS). III. To evaluate the safety and tolerability.

TERTIARY/EXPLORATORY OBJECTIVES:

I. To evaluate biomarkers of response to treatment and mechanisms of resistance with pretreatment and post-treatment bone marrow and blood samples with deoxyribonucleic acid (DNA) and ribonucleic acid (RNA) sequencing and immune profiling by flow cytometry.

OUTLINE:

Patients receive ixazomib orally (PO) on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab intravenously (IV) over 4-8 hours on days 1, 8, 15, and 22 of cycle 1. Beginning in cycle 3, patients receive rituximab IV over 4-8 hours on day 1. Treatment repeats every 28 days up to cycle 12 in the absence of disease progression or unacceptable toxicity. Patients benefiting from treatment may continue to receive ixazomib indefinitely in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of mantle cell lymphoma
* Patients must have measurable disease, as defined by at least one of the following:

  * Lymph node or mass 2 cm or greater, splenomegaly > 13 cm
  * Bone marrow only disease as per morphology or flow cytometry
* Patients must have relapsed and/or refractory disease to at least 2 lines of therapy including either an anthracycline- or bendamustine- based regimen and a BTK inhibitor
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelets >= 50,000/mm^3
* Total bilirubin < 1.5 x institutional upper limit of normal (ULN). In patients with documented Gilbert's syndrome, total bilirubin =< 2.5 x ULN
* Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) =< 3 x ULN
* Creatinine clearance >= 30 mL/min
* Patients must be willing to give written consent before performance of any study related procedures not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Failure to have fully recovered (i.e., =< grade 1 toxicity) from the reversible effects of prior chemotherapy
* Major surgery within 14 days before enrollment
* Radiotherapy within 14 days before enrollment. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib
* Central nervous system involvement
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment. Patient may be eligible, if infectious disease specialist approves start of therapy AND subject has completed course of antibiotic therapy
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort
* Ongoing or active systemic infection, active (deoxyribonucleic acid [DNA] polymerase chain reaction [PCR] positivity) hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Patient has >= grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination during the screening period
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial
* Patients that have previously been treated with proteasome inhibitors, or participated in a study with proteasome inhibitors whether treated with proteasome inhibitors or not

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hun J Lee, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open label, single center, single-arm, phase II
Groups:
- Study Drug: Ixazomib 4mg PO on days 1, 8, 15 Rituximab 375 mg/m2 IV weekly until cycle 3, then given day 1 of each cycle
Period: Overall Study
Arm/Group | Study Drug
Started | 3
Completed | 2
Not Completed | 1
Not completed — Progressive Disease | 1

BASELINE CHARACTERISTICS:
Population: Patients that received at least one dose of the study drug
Arm/Group | Study Drug
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants] — Patients that received at least one dose of study drug
  Participants
    <=18 years | 0
    Between 18 and 65 years | 1
    >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Patients that received at least one dose of the study drug
  Participants
    Female | 1
    Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Patients that received at least one dose of the study drug
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 2
    Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Patients that received at least one dose of the study drug
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 2
    More than one race | 0
    Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate at 16 Weeks
Description: Evaluate the complete remission rate of BTK inhibitor refractory MCL patients with ixazomib and rituximab at 16 weeks of therapy. Complete remission at 16 weeks was measured by PET/CT or CT imaging using Lugano Criteria 2014.
Time Frame: 16 weeks
Population: All endpoints will be measured on patients that received at least one dose of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: Overall Response Rate at 16 Weeks
Description: Evaluate the overall response rate (ORR) assessed by Lugano criteria (2014)
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug
Number analyzed (Participants) | 3
Participants | 3

3. Secondary Outcome: Progression Free Survival (PFS) and Overall Survival (OS)
Description: Evaluate progression free survival and overall survival
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug
Number analyzed (Participants) | 3
Participants
  Overall survival (OS) | 3
  Complete Metabolic Response (CMR) | 2

4. Secondary Outcome: Tolerability of Study Drug at Weeks 8, 16, 28, 42, and 56
Description: Tolerability of study drug at weeks 8, 16, 28, 42, and 56 using CTCAE v4.0 Toxicities or Adverse Events (grade 3 and up) were measured using CTCAE v 4.0 to determine the tolerability of ixazomib.
Time Frame: time of first dose of ixazomib through 30 days after the last dose of ixazomib was administered, up to 140 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug
Number analyzed (Participants) | 3
Participants
  Week 8 | 0
  Week 16 | 0
  Week 28 | 0
  Week 42 | 0
  Week 56 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after administration of the last dose of ixazomib, up to 140 weeks.
Description: Adverse event data collected using definitions from CTCAE v4.0
Arm/Group | Study Drug
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug (N=3)
Respiratory, thoracic, and mediastinal disorders- other, specify (COVID-19 pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug (N=3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Insomnia (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Nausea (General disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT04047797/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT04047797/ICF_001.pdf